CLINICAL TRIAL: NCT04828577
Title: Brain Network Modulation and Alcohol Use
Acronym: RP2B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Fralin Biomedical Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RP2B/22-016
Record Dates: First submitted 2021-03-26; First posted 2021-04-02 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol Use Disorder (AUD); rt-fMRI; behavioral economics
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Real Time Neurofeedback (Experimental): Real time neurofeedback will be based on a classifier of increasing or decreasing alcohol craving/demand fMRI patterns. Participants will try to modulate their brain patterns based on neurofeedback via a visual dial during an fMRI scan. Participants will be told they will be controlling the visual dial.
  Interventions: Behavioral: Real Time Neurofeedback

INTERVENTIONS:
Behavioral: Real Time Neurofeedback — Participants receive feedback from their own brain activity.

SUMMARY:
The investigators will use real-time fMRI neurofeedback to enhance participants' ability to control their ability to modulate alcohol valuation.

DETAILED DESCRIPTION:
All study procedures will take place during a single study visit. Before the imaging session, a research assistant will aid the participant to select salient images related to individualized future goals as well as alcohol images which elicit self-reported craving. All participants will complete two fMRI runs within a single session. In run 1 of the scan (offline classifier training), participants will perform an image viewing task displaying alternating blocks of these goal- and alcohol-related images. Between the image viewing blocks we will assess reinforcer pathology with brief in-scanner measures of alcohol valuation (BAAD). In total, there will be six blocks each of the goal-oriented images, alcohol-related images, and BAAD (18 blocks total). Since this is a proof-of-concept experiment, the interspersed BAAD blocks will enable monitoring and validating changes in the participant's alcohol valuation after the image viewing blocks. Only the fMRI measures of goal- and alcohol-related image viewing will be used to build a support vector classifier (SVC). The participants will see a dial with a needle on the screen along with instructions to think of either future goals or alcohol cues. The dial will be directly controlled by ongoing output from the SVC, updating the needle position as participants imagine immediate (alcohol-related) or delayed (goal-related) cues. Based on this, it is expected that participants will have increased whole-brain signal-to-noise for alcohol vs. goal fMRI analyses and increased recruitment of frontal-parietal networks from enhanced visual attention to the task.

ELIGIBILITY:
Inclusion Criteria:

* self-report alcohol abuse
* be 21 years of age or older
* have a desire to quit or cut down on their drinking, but do not have proximate plans to enroll in treatment for AUD during the study period

Exclusion Criteria:

* meeting moderate to severe DSM-5 criteria for substance-use disorders other than alcohol or nicotine
* having a current diagnosis of any psychotic disorder
* having a history of seizure disorders or traumatic brain injury
* having any contraindication for participation in the MRI sessions
* reporting current pregnancy or lactation

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M LaConte, PhD, Principal Investigator — Fralin Biomedical Research Institute (FBRI) at VTC; Warren K Bickel, PhD, Principal Investigator — Fralin Biomedical Research Institute (FBRI) at VTC
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will adhere to all NIH requirements regarding data sharing. Participant data collected in this project will be de-identified and made available on a shared secured data repository. We will also share the analysis results. As part of this process, all investigators will be required to agree to the following conditions: 1) will adhere to the reporting responsibilities; 2) will not redistribute the data beyond the requesting individual and named collaborators; 3) will give appropriate acknowledgement; 4) will not use the data for commercial purposes; and 5) will obtain appropriate ethical approvals. Results from research conducted will be shared and disseminated, including: regular project meetings, annual meetings, symposia, workshops, and/or conferences for related groups. Manuscripts will be written and submitted for publication in peer-reviewed journals/conferences, following the NIH Public Access Policy guidelines. All necessary ethical approvals will be obtained.
Time Frame: Data will be made available upon request after dissemination of results.
Access Criteria: Data requests will be reviewed by the principal investigator and data will be shared with the expectation of acknowledgment of funding source and primary study team.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real Time Neurofeedback
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Real Time Neurofeedback
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Neurofeedback Control
Description: Participants were asked to move a neurofeedback dial to "alcohol" or "goal" directions. For the "alcohol" they were instructed to attempt to crave alcohol, and for the "goal" they were instructed to attempt to project themselves into their future goals. The outcome was measured by the mean correlation of the needle movement compared to the instructed needle movement.
Time Frame: During the real time fMRI scan, approximately 1 hour (single session)
Measure: Mean (Standard Deviation); unit: correlation coefficient
Arm/Group | Real Time Neurofeedback
Number analyzed (Participants) | 21
correlation coefficient | 0.061 (0.190)

ADVERSE EVENTS:
Time Frame: During the real time fMRI scan, approximately 1 hour (single session)
Arm/Group | Real Time Neurofeedback
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT04828577/Prot_SAP_000.pdf